CLINICAL TRIAL: NCT06748352
Title: Safety and Efficacy of Traction Robot-assisted Endoscopic Submucosal Dissection for Early Gastric Cancer: a Pilot Randomized Controlled Study
Brief Title: Safety and Efficacy of Traction Robot-assisted Endoscopic Submucosal Dissection for Early Gastric Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Xiuli Zuo, Professor, MD, PhD, Shandong University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SDU-QILU-G015
Record Dates: First submitted 2024-12-17; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Early Gastric Cancer; Endoscopic Submucosal Dissection; Robot Surgery
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FASTER-assisted ESD group (Experimental): Patients in this group undergo ESD with the assistance of the FASTER system.
  Interventions: Procedure: FASTER-assisted ESD
- Conventional ESD group (Active Comparator): Patients in this group undergo ESD following the clinically established pattern.
  Interventions: Procedure: Conventional ESD

INTERVENTIONS:
Procedure: FASTER-assisted ESD — The patients who are randomly assigned to the FASTER-assisted ESD group will undergo the ESD procedure with the assistance of the FASTER system.
  Arms: FASTER-assisted ESD group
Procedure: Conventional ESD — The patients who are randomly assigned to the conventional ESD group will undergo the ESD following the clinically established pattern.
  Arms: Conventional ESD group

SUMMARY:
The goal of this clinical trial is to investigate whether the flexible auxiliary single-arm transluminal endoscopic robot (FASTER) system can improve the safety of the endoscopic submucosal dissection (ESD). It will also evaluate the efficacy of the system, such as whether it could reduce the procedure time and so on. The main questions it aims to answer are:

Does the use of the FASTER system reduce the number of muscular injuries, improving the safety of the ESD procedure? Does the use of the FASTER system reduce the procedure and dissection time, improving the efficacy of the ESD procedure? Researchers will compare FASTER-assisted ESD and conventional ESD to evaluate the safety and efficacy of the FASTER system.

Participants will:

Be randomly assigned to the group with ESD using the traditional procedure or to the group with ESD assisted by the FASTER system.

Keep a diary of their symptoms after the procedure. ESD has gained widespread acceptance as the standard method for treating early-stage gastrointestinal cancers. Adequate exposure of the submucosa layer through effective tissue traction is vital for the safe and effective performance of ESD. The FASTER system is designed to overcome this technical difficulty.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-80.
* Patients with pathologically verified high-grade intraepithelial neoplasia (HGIN) or intramucosal carcinoma of the stomach.

Exclusion Criteria:

* Patients have lesions with confirmed or potential deep submucosal invasion or lymph node metastasis.
* Patients with severe underlying diseases precluding endotracheal intubation, general anesthesia, or surgery.
* Patients have a history of gastric malignancy with previous radiotherapy or operative treatment leading to changes in gastric structure.
* Patients have lesions with local recurrence after endoscopic resection.
* Patients unable to obtain informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-12-30 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
the number of muscular injuries | Within 24 hours after the procedure.
  Muscular injury is described as visible damage to the muscularis propria.

SECONDARY OUTCOMES:
the incidence of muscular injury | Within 24 hours after the procedure.
  Muscular injury is described as visible damage to the muscularis propria.
the frequency of intraoperative hemorrhage | Within 24 hours after the procedure.
the proportion of intraoperative hemorrhage ≥ grade 2 | Within 24 hours after the procedure.
  Intraoperative hemorrhage is divided into four grades: Grade 0 means no significant bleeding is observed during the procedure. Grade 1 means minimal bleeding, which could stop spontaneously or be easily controlled by cauterization with a dual knife. Grade 2 refers to minor hemorrhage that requires multiple cauterizations with a dual knife or hemostatic forceps. Grade 3 indicates massive hemorrhage that requires multiple cauterizations with hemostatic forceps.
hemostasis time | Within 24 hours after the procedure.
  Hemostasis time referred to the time from the detection of submucosal bleeding until hemostasis was completed.
the frequency of supplemental injections | Within 24 hours after the procedure.
  Supplemental injection refers to injections performed after the beginning of the dissection.
the supplemental injections time | Within 24 hours after the procedure.
  The time of supplementary injection is from the insertion of the injection needle into the submucosal layer until the injection is completed and the needle is withdrawn.
procedure time | Within 24 hours after the procedure.
  Procedure time is the time from the beginning of injection to the completion of dissection.
dissection time | Within 24 hours after the procedure.
  Dissection time is the time from the beginning of dissection to the completion of dissection.
direct-vision dissection rate | Within 24 hours after the procedure.
  Direct-vision dissection time is the time that the endoscopist can directly observe the tip of the dual knife and the submucosal layer at the same time. By dividing the direct-vision dissection time by the total dissection duration, the direct-vision dissection rate is calculated.
en bloc resection rate | Within 24 hours after the procedure.
  En bloc dissection refers to the complete removal of the entire lesion in a single piece.
R0 resection rate | Within 24 hours after the procedure.
  R0 resection is defined as en bloc resection with negative vertical and horizontal margins.

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China